CLINICAL TRIAL: NCT04811547
Title: Adding Ankle Brachial Index to Traditional Framingham Risks Can Improve All-cause Mortality and Cardiac Mortality Prediction in Medium and High Framingham Risk Score Patients: A China Prediction Model
Brief Title: Ankle-Brachial Index to Predicte All-Cause and Cardiovascular Mortality in Framingham Risk Score Patients
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, cardiology department of shanghai 10th people's hospital, Shanghai 10th People's Hospital
Other Study IDs: AIRPORTS
Record Dates: First submitted 2021-03-13; First posted 2021-03-23 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-03

CONDITIONS: Ankle Brachial Index
Keywords: Atherosclerosis risk; Ankle Brachial Index; Framingham Risk Score; Prediction Model; All-cause Mortality; Cardiac Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ankle-Brachial Index value: Valid participants were separated into 0-0.60, 0.61-0.90, 0.91-0.99, and 1.00-1.40 four ABI subgroups.

SUMMARY:
Framingham Risk Score (FRS) included age, gender, body mass index (BMI), cigarette smoking, blood pressure, total cholesterol (TC), LDL-cholesterol (LDL-C) and diabetes mellitus (DM). Previously, Framingham cohort study and other study has confered patients with medium or high FRS had worse prognosis. However, the score list was tending to over-estimate risk in medium FRS or under-estimate risk in high FRS patients . For this reason, ACC/AHA cholesterol guidelines also recommend the use of additional markers to improve atherosclerotic cardiovascular disease (ASCVD) risk assessment and medical decision making.

Meanwhile, the ABI, which was the ratio of systolic pressure at the ankle to that in the arm, was quick, easy and used to diagnosis and assess the severity of peripheral artery disease (PAD) in the legs. Several research have shown its low value as an indicator of general atherosclerosis and independently risk associated with cardiovascular events in prospective studies . In addition, ABI aggressively modified risk factors and accelerated the adverse prognosis of ASCVD. However, whether FRS or ABI, were all related to participants and race. And, most studies were from western countries, lack of Asian date, especially aimed at risk prediction model research. Therefore, this research was aimed to validate incorporating ABI and relevant Framingham risk variables whether could improve prediction all-cause mortality and cardiac mortality in medium and high Framingham risk score (FRS) patients.

DETAILED DESCRIPTION:
The study is a longitudinal cohort study. The first cross-sectional survey was conducted in 2011.

ELIGIBILITY:
The inclusion criteria:

1. Patients were age older than or equal to 18 years
2. Patients with medium and high Framingham risk score，namely, Framingham Risk Score (FRS) 10%-20%,or FRS > 20%.
3. All participants gave written informed consent to this study, which was approved by the ethics committee of Tongji University.

Exclusion Criteria:

1. Patients were suffering from mental illness.
2. Life expectancy of patients were less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There were 3687 participants from multi-central departments with multiple classical Framingham risk factors atherosclerosis, including 1935 males and 1752 females whose age older than or equal to 18 years. All participants were followed up from November 2011 to June 2018. A total of hospitalized patients were consecutively enrolled from cardiology department and under treatment because of cardiovascular diseases .
Sampling Method: Probability Sample
Enrollment: 3687 (Actual)
Dates: Start 2011-11-20 (Actual); Primary Completion 2013-03-12 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
All-Causes mortality and Cardiac mortality | from November 2011 to June 2018
  In this study, the Cardiac death was only cardiac event death. Medical records and death certificates of all patients who had an event were obtained and validated by cardiologist. Death was confirmed from hospital records or by contact with participants and their families. All materials were reviewed independently by five senior physicians of the cohort study to confirm the cause of death.

SECONDARY OUTCOMES:
New-onset Cardiovascular Events | from November 2011 to June 2018
  New-onset Cardiovascular events are composed of cardiac including non-fatal myocardial infarction, unstable angina, and coronary revascularization procedures during follow-up time. Exclusion criteria were stale angina (>6 months), revascularization procedure for CAD ( >6 months) and myocardial infarction( >6 months).